CLINICAL TRIAL: NCT05768633
Title: Counterfactual Thinking About Clinical Decision and Decision-making in the Context of Obstructive Sleep Apnea Syndrome.
Brief Title: Counterfactual Thinking and Decision-making in OSA Syndrome
Acronym: CT_OSAS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C211
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: counterfactual thinking; decision-making; neuropsychological assessment; clinical setting
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Individuals diagnosed with obstructive sleep apnea (OSA) syndrome recruited at the beginning of rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy).
  Interventions: Behavioral: Counterfactual Inference Test
- Controls: Age-matched healthy individuals recruited outside the hospital through personal contacts of the researchers and word-of-mouth.
  Interventions: Behavioral: Counterfactual Inference Test

INTERVENTIONS:
Behavioral: Counterfactual Inference Test — All participants will be asked to complete the Counterfactual Inference Test - CIT (McNamara et al., 2003), a neuropsychological test that measures the ability to produce counterfactual-derived inferences. Moreover, the decision-making ability will be specifically tested through ad-hoc questionnaire (i.e., the Decision-Making Questionnaire). Finally, all participants will be screened with an extensive neuropsychological assessment, particularly on executive functioning.

SUMMARY:
The aim of this research is to verify the ability of counterfactual thinking about medical decisions in individuals with obstructive sleep apnea syndrome when compared with healthy individuals

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of obstructive sleep apnea syndrome, according to the clinical assessment.

Exclusion Criteria:

- Concurrent neurological, neurodevelopmental (e.g., autism), motor, and/or psychiatric disorders

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with obstructive sleep apnea syndrome consecutively recruited at the beginning of their rehabilitative treatment at the IRCCS Istituto Auxologico Italiano.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
CIT score | Baseline
  Score at the Counterfactual inference test (CIT). The questionnaire is a four question forced choice test based on past research regarding factors that enhance counterfactual thinking. For each of the four questions, events experienced by two individuals are presented, and three response options are given. Only one option is the valid: the score is 1. For the not valid options, the score will be 0. Overall, the score range for the questionnaire is from 0 (worse performance) to 4 (best performance).

SECONDARY OUTCOMES:
Decision-making index | Baseline
  Score at the Decision-Making Questionnaire. The self-report questionnaire assesses the decision making ability according to 7 questions, with a 5-item Likert's scale. The overall score (i.e., the sum of the scores at all questions) can range from 7 (worse decision making strategy) to 35 (best decision making strategy).

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Tagini, PhD, Principal Investigator — IRCCS Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy